CLINICAL TRIAL: NCT05410652
Title: A Multicenter Clinical Study of Helicobacter Pylori 23S rRNA/gyrA Gene Mutation Detection Kit (Fluorescence PCR Fusion Curve Method)
Brief Title: Helicobacter Pylori 23S rRNA/gyrA Gene Mutation Detection Kit (Fluorescence PCR Fusion Curve Method)
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Senior professional title, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: QX202200516-01
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Helicobacter Pylori Infection; Helicobacter Pylori gyrA Levofloxacin Resistance Mutation; Fecal Drug Resistance Gene Detection; Helicobacter Pylori Infection, Susceptibility to
Keywords: Fecal gene detection; Levofloxacin resistance gene; Clarithromycin resistance gene

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fecal kit group: Collect stool samples from patients who meet the inclusion criteria. DNA was extracted from fecal samples. After that, the extracted DNA was sequenced by first generation sequencing. Finally，the mutation sites of extracted DNA were detected by fecal gene detection kit.
  Interventions: Diagnostic Test: Detection of fecal samples with diagnostic kit
- Sanger Sequencing group: Detection of gyrA and 23S rRNA mutations in H. pylori isolated from Gastric Mucosa by Sanger Sequencing
  Interventions: Diagnostic Test: Sanger Sequencing group
- Drug sensitivity test group: Gastroscopy was performed on patients who met the inclusion and exclusion criteria to obtain samples of gastric mucosa. Helicobacter pylori culture and drug sensitivity test were performed on gastric mucosa samples in vitro. Finally, the drug sensitivity test results were collected.
  Interventions: Diagnostic Test: Bacterial culture and drug sensitivity test of gastric mucosa samples

INTERVENTIONS:
Diagnostic Test: Detection of fecal samples with diagnostic kit — The 23S rRNA mutation site of clarithromycin and gyrA mutation site of levofloxacin were detected by Helicobacter Pylori fecal Gene Mutation Detection Kit.
  Groups: Fecal kit group
Diagnostic Test: Sanger Sequencing group — Detection of gyrA and 23S rRNA mutations in H. pylori isolated from Gastric Mucosa by Sanger Sequencing
  Groups: Sanger Sequencing group
Diagnostic Test: Bacterial culture and drug sensitivity test of gastric mucosa samples — First, a sample of the patient's gastric mucosa will be obtained through gastroscopy. Then, Helicobacter pylori culture and drug sensitivity test can be carried out. Finally, the resistance data of Helicobacter pylori to clarithromycin and levofloxacin will be obtained.
  Groups: Drug sensitivity test group

SUMMARY:
The purpose of this study was to evaluate the detection ability of Helicobacter pylori 23S rRNA/gyrA gene mutation detection kit (fluorescent PCR fusion curve method) for Helicobacter pylori gene mutation.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requriment will be included in this simultaneous blind test.

ELIGIBILITY:
Inclusion Criteria:

* 1. patients with Helicobacter pylori infection who need gastroscopy; 2. patients with positive Helicobacter pylori culture in gastric mucosa 3. Helicobacter pylori negative patients

Exclusion Criteria:

* 1.Patients with insufficient fecal samples collected 2.Patients with contraindication of gastroscopic biopsy

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will collect patients aged 18-70 years with or without Helicobacter pylori infection who have the need for gastroscopy.
Sampling Method: Probability Sample
Enrollment: 1176 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of consistency between fecal gene detection kit and Drug sensitivity test | 4 weeks
  Compare the positive coincidence rate, negative coincidence rate, total coincidence rate and consistency between stool gene detection kit and drug sensitivity test
Evaluation of consistency between fecal gene detection kit and first generation sequencing | 4 weeks
  Compare the positive coincidence rate, negative coincidence rate, total coincidence rate and consistency between stool gene detection kit and first generation sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Zhang, Master, Study Chair — Nanjing First Hospital, Nanjing Medical University; Yong Xie, Docter, Study Director — The First Affiliated Hospital of Nanchang University; Bin lv, Master, Study Director — The First Affiliated Hospital of Zhejiang Chinese Medical University; Bin Yang, Doctor, Principal Investigator — Jiangsu Taizhou People's Hospital
Locations (4):
- China (4):
  - Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Jiangsu Taizhou People's Hospital, Taizhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei WJ, He BS, Lv B, Yang B, Xie Y, Zhang ZY. Clinical evaluation of a novel H. pylori fecal molecular diagnosis kit (multiplex RT-PCR method) for detecting clarithromycin and fluoroquinolones resistance using stool samples. Front Cell Infect Microbiol. 2025 Jun 23;15:1592612. doi: 10.3389/fcimb.2025.1592612. eCollection 2025. PMID 40625832